CLINICAL TRIAL: NCT01204866
Title: A Phase I, Open Label, Controlled Study of Valortim® (MDX-1303) and Its Selected Formulation Components When Introduced Percutaneously in Subjects Who Have and Have Not Been Exposed to Valortim Administered Intravenously
Brief Title: Study of Valortim® (MDX-1303) and Its Selected Formulation Components Percutaneous Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmAthene, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Pharmathene, Inc., Clinical Project Manager
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0036-08-05-A; HHSN272200700033C (Other Grant/Funding Number: BAA-NIH-NIAID-DMID-07-37); 09-0117 (Other Grant/Funding Number: HHSN272200700033C)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Allergic Reactions
Keywords: Allergic-Like Reaction; Selected Formulation Components
MeSH Terms: conditions — Hypersensitivity | interventions — Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stage I (Experimental): Three (3) healthy male or female volunteers aged 18-59 years, not previously exposed to Valortim and who do not have pre-existing allergies
  Interventions: Biological: Valortim and selected Components
- Stage II (Experimental): Up to 4 healthy male or female volunteers aged 18-59 previously exposed to intravenous (IV) Valortim in PharmAthene Study #0036-08-05
  Interventions: Drug: Valortim and Selected Components

INTERVENTIONS:
Biological: Valortim and selected Components — * Valortim (Lot #10-08-001, 25 mg/mL) will be filtered through a 0.22 µm syringe filter and diluted 1:1000, 1:100, 1:10, and 1:1 in saline.
  * Polysorbate 80 will be diluted in saline to the following concentrations: 0.06 mg/mL, 0.2 mg/mL, and 0.6 mg/mL.
  * Mannitol (30 mg/mL) will be diluted in saline to the following concentrations: 1:1000, 1:100, 1:10, and 1:1
  * Histamine (1 mg/mL), positive control
  * Saline (0.9%), negative control
  Other Names: Anthrax
  Arms: Stage I
Drug: Valortim and Selected Components — • It is anticipated that up to 4 subjects that received Valortim in a previous study (#0036-08-05) will participate in Stage II of the study; two of these subjects experienced adverse events while being dosed with Valortim. Subjects will each be tested percutaneously with Valortim, polysorbate 80, mannitol, histamine, and saline.
  * Only one subject will be skin tested in a single day.
  * The appropriate dilution for Valortim, mannitol, and polysorbate 80 will be based on the results from Stage I of this study. As was done in Stage I, Valortim will be filtered through a 0.22 µm syringe filter. Histamine (1 mg/mL) and saline (0.9%) will be used as the positive and negative controls, respectively
  Other Names: Anthrax
  Arms: Stage II

SUMMARY:
The purpose of this study is to determine if Valortim, or one or more of its selected formulation components, induces a wheal reaction when introduced percutaneously.

Two of 4 subjects dosed in a previous study with a modified formulation of Valortim experienced treatment related adverse events which were suggestive of allergic or allergic-like reactions. In order to better characterize these reactions and determine if they represent allergic or allergic-like reactions to Valortim or one or more of its components, skin testing of Valortim and selected components on naïve and Valortim-exposed subjects will be performed in this study

DETAILED DESCRIPTION:
A maximum of 7 subjects will participate in the study. Up to four of these subjects have been previously exposed to IV Valortim.

The study will be conducted in two stages. The first stage will be performed on subjects not previously exposed to Valortim (Valortim-naïve subjects), to determine the correct dilutions of the test components. The second stage will be performed on the Valortim-exposed subjects using the dilutions of test components as determined in the first stage of the study.

The following components will be tested to determine their ability to induce a wheal reaction shortly after exposure to the skin by percutaneous application by needle prick: Valortim (Lot# 10-08-001), polysorbate 80, mannitol, histamine (positive control), and saline (negative control). All components except histamine will be provided to the clinical site by PharmAthene with detailed instructions for handling, storage, and dilution. A tiny drop of the aforementioned components will be introduced onto the surface of the skin and the skin will be pricked, allowing the components to enter the surface of the skin. Multiple components will be tested on the subjects' forearms or back; location of testing to be determined by scars, moles,pre-existing skin lesions, or other issues deemed by the Principal Investigator (PI) to have the potential to interfere with interpretation of the results.

Stage I:

* 3 Valortim-naïve, non-allergic subjects
* Only one subject will be skin tested in a single day
* Subjects will be tested percutaneously with the above mentioned components at the following dilutions:

  * Valortim (Lot #10-08-001, 25 mg/mL) will be filtered through a 0.22 µm syringe filter and diluted 1:1000, 1:100, 1:10, and 1:1 in saline.
  * Polysorbate 80 will be diluted in saline to the following concentrations: 0.06 mg/mL, 0.2 mg/mL, and 0.6 mg/mL.
  * Mannitol (30 mg/mL) will be diluted in saline to the following concentrations: 1:1000, 1:100, 1:10, and 1:1
  * Histamine (1 mg/mL), positive control
  * Saline (0.9%), negative control.
* Multiple dilutions of Valortim, polysorbate 80, and mannitol will be used to determine the appropriate dilution for the second stage of the study in an attempt to avoid the possibility of a false positive reaction due to irritation.
* The starting dilution for Valortim and mannitol will be 1:1000 and will move progressively to more concentrated dilutions (1:100, 1:10, 1:1). The starting dilution for polysorbate 80 will be 0.06 mg/mL and will also move progressively higher to concentrations of 0.2 mg/mL and 0.6 mg/mL respectively.
* Fifteen minutes after the application of the test articles, the skin test sites will be examined for a wheal reaction. The skin sites will be examined again 1 hour following testing, just prior to discharge from the clinic. Subjects will return at 1 and 2 days following testing to assess the skin testing sites and to observe for any adverse events.
* A skin test is considered positive if, at 15 minutes following application, the wheal produced by the test article is equal to or greater than, that caused by positive control (histamine), or is at least 3 mm greater than the wheal of negative control (saline).
* A negative skin test is no wheal, or a wheal less than 3 mm larger than the saline control as determined at 15 minutes following application.

Stage II:

* It is anticipated that up to 4 subjects that received Valortim in a previous study (#0036-08-05) will participate in Stage II of the study; two of these subjects experienced adverse events while being dosed with Valortim. Subjects will each be tested percutaneously with Valortim, polysorbate 80, mannitol, histamine, and saline.

  * Only one subject will be skin tested in a single day.
  * The appropriate dilution for Valortim, mannitol, and polysorbate 80 will be based on the results from Stage I of this study. As was done in Stage I, Valortim will be filtered through a 0.22 µm syringe filter. Histamine (1 mg/mL) and saline (0.9%) will be used as the positive and negative controls, respectively.
* Fifteen minutes after the application of the test articles and pricking the skin, the skin test sites will be examined for a wheal reaction. The skin sites will be examined again 1 hour following testing, just prior to discharge from the clinic. Subjects will return at 1 and 2 days following testing to assess the skin testing site and to observe for any adverse events.
* A skin test is considered positive if the wheal produced by the test article 15 minutes following application is equal to or greater than that caused by positive control (histamine), or is at least 3 mm greater than the wheal of negative control (saline).
* A negative skin test is no wheal, or a wheal less than 3 mm larger than the saline control as determined at 15 minutes following application.

ELIGIBILITY:
Inclusion Criteria:Stage I Subjects

* In the opinion of the Investigator, subjects should be in generally good health, based upon pre-study medical history and abbreviated physical exam.
* Female subjects cannot be pregnant, as confirmed by a negative urine pregnancy test at Study Day 1, prior to skin testing.
* Women of childbearing potential may be enrolled if one of the following criteria applies:

  * Must be using an effective form of contraception for at least one month prior to study entry, must have a negative urine pregnancy test on Day 1, prior to skin testing
  * Is sexually abstinent
  * Is monogamous with a vasectomized partner (>3 months prior)
  * Is postmenopausal (i.e. no cycle for at least the previous 12 months, is of menopausal age (>45 years) and has a negative urine pregnancy test on Day 1, prior to skin testing
  * Is surgically sterilized
  * Has had a total hysterectomy
* Sexually active male subjects may be enrolled if one of the following criteria applies:

  * Has had a vasectomy
  * Using condoms and whose partner is using an acceptable form of contraception *Is sexually abstinent.
* In addition to the Inclusion Criteria above, Stage II Subjects must also meet the following criteria :

  * Must have participated in PharmAthene Study #0036-08-05 and have been previously exposed in that study to Valortim.

Exclusion Criteria: Stage I & II

* Antihistamine use within 14 days of testing. Medications with antihistamine properties (i.e., anticholinergic agents, phenothiazine), beta-blockers, MAO-inhibitors or tricyclic antidepressant use within 1 day of testing.
* Dermatographia, or extreme skin sensitivity.
* History of allergic rhinitis, asthma or eczema.
* Outward signs of active allergies or upper respiratory infection.
* Known pregnancy as confirmed by urine pregnancy testing on Day 1, prior to skin testing procedures.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Skin Testing Results | Initial results assessed after 15minutes and up to 72 hours.
  Assessment of any wheal reaction from the study drug or its selected components and how this compares to the positive and negative control

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wald, MD, Principal Investigator — Kansas City Allergy and Asthma; Valerie Riddle, MD, Study Director — Sponsor Medical Monitor
Locations (1):
- Kansas City Allergy and Asthma, Overland Park, Kansas, United States